CLINICAL TRIAL: NCT02414074
Title: Adaptive Intervention Strategies in Conduct Problems Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); St. Paul Youth Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1304S30941; R34MH097832 (NIH)
Record Dates: First submitted 2015-04-03; First posted 2015-04-10 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Conduct Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Youth Behavioral Intervention (Other): Teen Intervene Program
  Interventions: Behavioral: Youth Behavioral Intervention
- Parent Education (Other): Everyday Parenting Program
  Interventions: Behavioral: Parent Education

INTERVENTIONS:
Behavioral: Youth Behavioral Intervention — Teen Intervene is an early intervention program for 12-19 year olds.
  Other Names: Teen Intervene
  Arms: Youth Behavioral Intervention
Behavioral: Parent Education — Everyday Parenting is a parent training curriculum.
  Other Names: Everyday Parenting
  Arms: Parent Education

SUMMARY:
This pilot study conducts feasibility research to develop adaptive intervention strategies for conduct problems prevention. The adaptive model will stipulate for whom only brief prevention strategies are sufficient and for whom more intensive strategies are necessary. The research will involve youth (10-17 years of age) identified by law enforcement as early offenders and who are referred for pre-court juvenile diversion programming.

DETAILED DESCRIPTION:
This project proposes to conduct feasibility research to inform implementation of a future full-scale SMART design (i.e., sequential, multiple assignment, randomized trial) that will be used to construct adaptive intervention strategies (AIS) for conduct problems prevention. AIS individualize treatment via decision rules that specify how the type (youth-focused or parent focused) or intensity (low dosage or high dosage) of an intervention should be formulated prior to the beginning of treatment based on youth and family characteristics and/or repeatedly adjusted over time based on proximal outcomes collected during treatment. AIS are needed in conduct problems prevention to address the heterogeneity of at-risk youth and the variability in response to conventional fixed-type preventive interventions. With the present SMART trial each participant will progress through two stages of intervention using a stepped-care framework. In the first stage participants will be randomized to one of two 'brief-type' intervention options, either the youth-focused Teen Intervene-Brief program (TI-B; Winters & Leitten, 2007) or the parent-focused Everyday Parenting-Brief program (EP-B; Dishion et al., 2003, 2010). Responders to either program will be stepped down and monitored over time for maintenance. Non-responders to either program will be stepped up and randomized to one of two second stage 'intensive-type' intervention options that feature either (1) continuation of the first stage option with increased dosage (EP-Expanded or TI-Expanded), or (2) switching to the alternative expanded intervention modality. This feasibility study will enroll high risk youth (10-17 years of age) who have been arrested for status or misdemeanor offenses and referred for pre-court juvenile diversion programming. The aims of this feasibility research are to (1) develop practice infrastructure for implementing a SMART design and assess practitioner adherence to the various intervention sequences, (2) roll out the stepped-care intervention sequences and obtain estimates of recruitment into SMART, attrition at both stages, and overall response rate to first-stage intervention options, (3) describe the demographic and clinical characteristics of the sample of diversion-referred youth who are enrolled in the study, (4) create a latent construct for conduct problems that will be used as the distal outcome, and (5) explore the utility of incorporating secondary tailoring variables (e.g., child and family risk characteristics) in the adaptive intervention model.

ELIGIBILITY:
Inclusion Criteria:

* Youth ages 10-17
* Juvenile diversion referral (to community partner agency)

Exclusion Criteria:

* Pervasive developmental disabilities
* Serious psychiatric disorders requiring specialized mental health treatment (e.g. psychosis, bipolar disorder, etc.)
* Substance dependence

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Peer Delinquency Scale | 9 months
  Youth Report
Family Check-Up Youth Questionnaire - Adolescent | 9 months
  Youth Report
Personal Experiences Screening Questionnaire-Adolescent | 9 months
  Youth Report
Self-Reported Delinquency Scale-Adolescent (SRD) | 9 months
  Youth Report
Inventory of Callous-Unemotional Traits-Youth (ICU) | 9 months
  Youth Report
Delayed Discounting Task | 9 months
  Youth Computer Task
Dimensional Change Card Sort Task (DCCS) | 9 months
  Youth Computer Task
Flanker Task | 9 months
  Youth Computer Task
Iowa Gambling Task | 9 months
  Youth Computer Task
Family Check-Up Caregiver Questionnaire-Adolescent | 9 months
  Parent Report
Behavior Assessment System for Children (BASC-2) | 9 months
  Parent Report
Delis Rating of Executive Functions (D-REF) | 9 months
  Parent Report
Family Check-Up Caregiver Questionnaire-Family | 9 months
  Parent Report
Early Adolescent Temperament Questionnaire-Revised (EAT-Q) | 9 months
  Parent Report
Disruptive Behavior Rating Scale (DBRS) | 9 months
  Parent Report
Parenting Relationship Questionnaire (PRQ) | 9 months
  Parent Report
Inventory of Callous-Unemotional Traits-Parent (ICU) | 9 months
  Parent Report

CONTACTS AND LOCATIONS:
Overall Officials: Gerald August, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- Center for Personalized Prevention Research in Children's Mental Health, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No